CLINICAL TRIAL: NCT00399984
Title: Enhancing Pediatric Asthma Management
Brief Title: Evaluating a Pediatric Asthma Management Education Program for Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 437; R01HL070771 (NIH)
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Asthma; Education, Medical
Keywords: Continuing Medical Education
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Asthma Education Program
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: Asthma Education Program — interactive seminars regarding daily inhaled corticosteroids
  Arms: 1

SUMMARY:
Inhaled corticosteroids taken on a daily basis have been proven to be the most effective treatment for children with persistent asthma. However, many pediatricians still do not prescribe daily corticosteroids to their asthmatic patients; this can lead to poor health outcomes among asthmatic children. This study will evaluate an interactive medical education program that focuses on improving pediatricians' asthma management skills and on encouraging increased corticosteroid use among their patients with asthma.

DETAILED DESCRIPTION:
Asthma is a common childhood disease that affects over 9 million children in the United States. In 1997, the National Heart, Lung, and Blood Institute (NHLBI) published a set of guidelines aimed at improving the quality of patient care for individuals with asthma. According to the guidelines, a daily dose of inhaled corticosteroids is considered the most effective treatment for the long-term control of asthma. Despite this recommendation, many pediatricians are not prescribing daily corticosteroids to asthmatic children who may benefit from this treatment.

Continuing medical education (CME) is viewed as the primary method of keeping health care providers informed of new research knowledge and the latest medical trends. While traditional CME programs have not been successful in changing physician behavior, an interactive program that offers skills development for implementing changes in the care and treatment of asthmatic patients may prove effective. The purpose of this study is to develop, implement, and evaluate an interactive asthma education program targeted towards pediatricians. Specifically, the study will determine the program's effectiveness at developing asthma management skills in pediatricians, including corticosteroid prescribing practices, and improving asthma-related outcomes among their pediatric patients.

In this 5-year study, pediatricians will be randomly assigned to either an asthma education intervention group or a control group. The intervention group will attend the enhanced asthma education seminar, and the control group will attend a traditional lecture about asthma. In Years 1 and 2, the intervention group will participate in a 2-hour focus group to discuss barriers to adopting the NHLBI asthma guidelines for daily corticosteroid therapy. A brief survey on this same topic will also be completed. During Year 2, physicians in the intervention group will attend at least 5 hours of educational seminars designed to improve adherence to the recommended guidelines. In Years 2 through 5, all physicians will complete yearly questionnaires to assess barriers to corticosteroid prescription methods. Parents of asthmatic patients treated by the pediatricians will take part in a 20-minute telephone survey each year, and study researchers will review the medical records of each child.

ELIGIBILITY:
Inclusion Criteria:

* Pediatricians must meet all of the following criteria:

  1. Graduate of a pediatric residency program in the United States
  2. In active medical practice for at least 4 half-day sessions, with 40% clinical effort in general pediatrics
  3. At least 54 children with asthma in their patient population
* Parents of pediatric asthma patients must meet all of the following criteria:

  1. Parent or guardian of a pediatric patient that meets patient eligibility criteria
  2. Able to identify that the participating physician is the child's primary care pediatrician
  3. Provides most asthma management or is the adult who normally takes the child to the doctor
* Pediatric patients must meet all of the following criteria:

  1. Older than 4 years of age (to decrease the likelihood that the child has bronchiolitis)
  2. Younger than 16 years of age (to ensure that during all 3 years of the evaluation part of the study, the child will be younger than 20 years of age)
  3. Diagnosis of asthma made by a physician using commonly accepted clinical criteria
  4. No other chronic disorders that have pulmonary complications (e.g., sickle cell disease, tuberculosis, acquired immune deficiency syndrome [AIDS], cystic fibrosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Changes in physician knowledge, attitudes, and self-reported behavior | 1-3 years
Changes in patient asthma outcomes (both measured on a yearly basis) | 1-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Cabana, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States